CLINICAL TRIAL: NCT01505647
Title: A Phase III Double-Blinded, Randomized, Multicenter, Controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of ZOSTAVAX™ Made With an Alternative Manufacturing Process (AMP)
Brief Title: Safety and Immunogenicity of Zoster Vaccine (ZOSTAVAX™) Made With an Alternative Manufacturing Process (AMP) (V211-042 AM1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V211-042
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Results first posted 2013-07-03 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Herpes Zoster; Shingles
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine; Adenosine Monophosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZOSTAVAX™ (AMP) (Experimental): ZOSTAVAX™ manufactured with an alternative process
  Interventions: Biological: Zoster Vaccine, Live (AMP)
- ZOSTAVAX™ (Active Comparator): ZOSTAVAX™ manufactured with the current process
  Interventions: Biological: Zoster Vaccine, Live

INTERVENTIONS:
Biological: Zoster Vaccine, Live (AMP) — One approximately 0.65-mL injection subcutaneously on Day 1
  Arms: ZOSTAVAX™ (AMP)
Biological: Zoster Vaccine, Live — One approximately 0.65-mL injection subcutaneously on Day 1
  Other Names: ZOSTAVAX™; V211
  Arms: ZOSTAVAX™

SUMMARY:
This study will determine whether ZOSTAVAX™ made with an alternative manufacturing process [ZOSTAVAX™ (AMP)] is well tolerated and immunogenic, and has a comparable immune response to ZOSTAVAX™.

ELIGIBILITY:
Inclusion Criteria:

* No fever on day of vaccination
* History of varicella or residence in a VZV-endemic area for ≥30 years
* Females of reproductive potential must have a negative pregnancy test and must agree to use acceptable methods of birth control

Exclusion Criteria:

* History of hypersensitivity reaction to any vaccine component
* Prior receipt of any varicella or zoster vaccine
* Prior history of herpes zoster
* Have recently had another vaccination
* Pregnant or breastfeeding
* Use of immunosuppressive therapy
* Known or suspected immune dysfunction
* Concomitant antiviral therapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2012-04; Primary Completion 2012-07 (Actual); Study Completion 2012-11 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] de Oliveira Gomes J, Gagliardi AM, Andriolo BN, Torloni MR, Andriolo RB, Puga MEDS, Canteiro Cruz E. Vaccines for preventing herpes zoster in older adults. Cochrane Database Syst Rev. 2023 Oct 2;10(10):CD008858. doi: 10.1002/14651858.CD008858.pub5. PMID 37781954

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant in the ZOSTAVAX™ (AMP) group was randomized but not vaccinated, making the number of participants vaccinated in this group 331
Groups:
- ZOSTAVAX™ (AMP): Zoster Vaccine, Live Alternative Manufacturing Process (AMP) : One approximately 0.65-mL injection subcutaneously on Day 1
- ZOSTAVAX™: Zoster Vaccine, Live : One approximately 0.65-mL injection subcutaneously on Day 1
Period: Day 1 Through Day 42 Follow-up
Arm/Group | ZOSTAVAX™ (AMP) | ZOSTAVAX™
Started | 332 | 166
Vaccinated | 331 | 166
Completed | 329 | 166
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Day 43 Through Day 182 Follow-up
Arm/Group | ZOSTAVAX™ (AMP) | ZOSTAVAX™
Started | 329 | 166
Completed | 328 | 163
Not Completed | 1 | 3
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- ZOSTAVAX™ (AMP): Zoster Vaccine, Live (AMP) : One approximately 0.65-mL injection subcutaneously on Day 1
- Total: Total of all reporting groups
Arm/Group | ZOSTAVAX™ (AMP) | ZOSTAVAX™ | Total
Number analyzed (Participants) | 332 | 166 | 498
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (7.1) | 62.4 (7.0) | 62.8 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 99 | 295
  Male | 136 | 67 | 203

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) of Varicella-Zoster Virus (VZV) Antibody
Description: VZV antibody titers were determined by glycoprotein enzyme-linked immunosorbent assay (gpELISA)
Time Frame: Day 1 and Week 6 postvaccination
Population: Analysis included all vaccinated participants except those who had protocol deviations that interfered with the assessment of antibody response, developed suspected varicella or herpes zoster rashes before blood sampling, or reported an exposure to varicella or herpes zoster
Measure: Geometric Mean (95% Confidence Interval); unit: Units/mL
Arm/Group | ZOSTAVAX™ (AMP) | ZOSTAVAX™
Number analyzed (Participants) | 330 | 166
Units/mL
  Day 1 postvaccination; n = 330, 166 | 235.7 [211.7 to 262.5] | 208.2 [176.4 to 245.7]
  Week 6 postvaccination; n = 320, 164 | 532.6 [489.2 to 579.9] | 457.1 [403.3 to 518.0]
Statistical Analysis 1: Comparison: ZOSTAVAX™ (AMP) vs ZOSTAVAX™; The hypothesis tested is that the GMT at Week 6 postvaccination with ZOSTAVAX™ (AMP) vaccine is non-inferior to that with the current process vaccine; Test type: Non-Inferiority or Equivalence — The GMT induced by ZOSTAVAX™ (AMP) vaccine is statistically non-inferior to that induced by the current process vaccine if the lower bound of the 95% confidence interval of the GMT ratio is >0.67; p < 0.001, Longitudinal regression model — The threshold for statistical significance is 0.025 (1-sided). The P-value was not adjusted; The analyzed GMT ratio, 95% confidence interval, and P-value were based on a longitudinal regression model adjusting for age and vaccination group; GMT Ratio = 1.08, 95% CI 2-sided [0.98 to 1.20]

2. Primary Outcome: Geometric Mean Fold Rise (GMFR) in VZV Antibody Titers
Description: VZV antibody titers were determined by gpELISA. The GMFR reports the geometric mean of the ratio of individual participant VZV antibody titers at Week 6 / Day 1 (Baseline).
Time Frame: Day 1 (Baseline) to Week 6 postvaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ZOSTAVAX™ (AMP) | ZOSTAVAX™
Number analyzed (Participants) | 320 | 164
Ratio | 2.3 [2.1 to 2.4] | 2.2 [2.0 to 2.5]
Statistical Analysis 1: Comparison: ZOSTAVAX™ (AMP); The hypothesis tested was that ZOSTAVAX™ (AMP) induces an acceptable GMFR in VZV antibody titer from prevaccination to 6 weeks postvaccination; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — The threshold for statistical significance is 0.025 (1-sided). The P-value was not adjusted

3. Secondary Outcome: Number of Participants With One or More Adverse Experiences (AEs)
Description: An AE is defined as any unfavorable and unintended change in the
  structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an adverse experience.
Time Frame: Day 1 to Day 42 postvaccination
Population: Analysis included all vaccinated participants with safety follow-up data. One participant in the AMP vaccine group was vaccinated but lost to follow-up without safety follow-up.
Measure: Number; unit: Participants
Arm/Group | ZOSTAVAX™ (AMP) | ZOSTAVAX™
Number analyzed (Participants) | 330 | 166
Participants | 205 | 99

4. Secondary Outcome: Number of Participants With One or More Serious Adverse Experience (SAE) Day 1 to 42 Postvaccination
Description: An SAE is defined as any adverse event that results in death, is life threatening, results in a persistent or significant disability/incapacity, results in hospitalization or prolongs an existing hospitalization, is a congenital anomaly/birth defect, is a cancer, is an overdose, or is considered an "other important medical event" based on medical judgement
Time Frame: Day 1 to Day 42 postvaccination
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | ZOSTAVAX™ (AMP) | ZOSTAVAX™
Number analyzed (Participants) | 330 | 166
Participants | 1 | 2

5. Secondary Outcome: Number of Participants With One or More Serious Adverse Experience Day 1 to 182 Postvaccination
Description: as for outcome 4
Time Frame: Day 1 to Day 182 postvaccination
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | ZOSTAVAX™ (AMP) | ZOSTAVAX™
Number analyzed (Participants) | 330 | 166
Participants | 4 | 8

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: Day 1 to Day 182 postvaccination; Other Adverse Events: Day 1 to Day 42 postvaccination
Arm/Group | ZOSTAVAX™ (AMP) | ZOSTAVAX™
Serious Adverse Events (participants affected / at risk) | 4/330 | 8/166
Other Adverse Events (participants affected / at risk) | 186/330 | 85/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZOSTAVAX™ (AMP) (N=330) | ZOSTAVAX™ (N=166)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Acquired oesophageal web (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder perforation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZOSTAVAX™ (AMP) (N=330) | ZOSTAVAX™ (N=166)
Injection-site erythema (General disorders) | 135 (138) | 66 (68)
Injection-site pain (General disorders) | 146 (153) | 68 (69)
Injection-site pruritus (General disorders) | 22 (23) | 13 (15)
Injection-site swelling (General disorders) | 106 (107) | 53 (56)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.